CLINICAL TRIAL: NCT01545466
Title: Mindfulness Based Stress Reduction for Adults With Migraines: A Pilot Study
Brief Title: Non-drug Interventions for Migraines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Rebecca Wells, Instructor, Brigham and Women's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011P001654
Record Dates: First submitted 2012-02-24; First posted 2012-03-06 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Migraine; Headache
Keywords: Migraines; Behavioral; Complementary and Alternative Medicine; Mindfulness Meditation; Mindfulness Based Stress Reduction
MeSH Terms: conditions — Migraine Disorders; Headache; Behavior | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Based Stress Reduction (Experimental): Participants will complete an 8 week course in Mindfulness Based Stress Reduction (MBSR), meeting once/week for 8 weeks and having a 4-6 hour retreat after the 6th class
  Interventions: Behavioral: Mindfulness Based Stress Reduction (MBSR)
- Wait-List Control Group (No Intervention): These participants will continue in usual care during the trial and will be offered the intervention of MBSR after the trial is over.

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction (MBSR) — MBSR involves 8 weekly 2 hour classes and one 4-6 hour retreat after the 6th class
  Arms: Mindfulness Based Stress Reduction

SUMMARY:
This proposal describes a randomized controlled pilot trial investigating feasibility, safety, and migraine frequency in patients with migraines who undergo an 8 week mindfulness based stress reduction (MBSR) program compared to a wait-list control group.

DETAILED DESCRIPTION:
Preliminary research has shown MBSR to be effective in chronic pain syndromes and other mind/body interventions have shown good promise in the treatment of headaches. A randomized controlled trial (RCT) of yoga in migraine without aura patients by John and colleagues showed that yoga resulted in a significant decrease in headache frequency, pain index, and symptomatic medication usage compared to a self-care group. This RCT demonstrated that patients with headaches may benefit from a mind-body intervention. However, their yoga protocol was not specified, and participants were instructed to practice the technique only during the prodromal phase of a headache (prior to the pain becoming severe), so as an abortive intervention at the time of a headache. Thus, the investigators of this trial are proposing to evaluate the effect of MBSR on adults with migraines compared to an education control group. This study will add to the John study because, unlike many other mind-body interventions, MBSR offers the distinct advantage of a standardized protocol that has been used both clinically and in numerous research studies across a wide variety of conditions. Furthermore, MBSR teaches participants a daily practice that, if effective, could serve as a prophylactic intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine (International Classification of Headache Disorders-II);21
* 4-14 days with migraines/month
* ≥one year of migraines
* ≥18 years
* Able and willing to attend weekly sessions and willing to participate in daily mindfulness assignments, up to 30-45 min/day
* Agreeable to participate and to be randomized to either group
* Fluent in English (since the treatment groups will be run in English)
* Good general health with no additional diseases expected to interfere with the study

Exclusion Criteria:

* Current regular meditation/yoga practice
* Any major systemic illness or unstable medical or psychiatric condition (e.g. suicide risk) requiring immediate treatment or that could lead to difficulty complying with the protocol
* Diagnosis of medication overuse headache (International Classification of Headache Disorders-II);19
* Current or planned pregnancy or breastfeeding
* New prophylactic migraine medicine started within 4 weeks of the screening visit
* Unwilling to maintain stable current doses of migraine medicines for the duration of trial
* Failure to complete baseline diary recordings of migraine activity and medication use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in Migraine frequency from Baseline | baseline, immediately post-intervention, 4 weeks post-intervention
  Change in the number of migraines per month from baseline(tracked with headache logs)

SECONDARY OUTCOMES:
Change in self-efficacy from baseline | baseline, immediately post-intervention, 4 weeks post-intervention
  Change in self-efficacy from baseline(Headache Management Self-Efficacy Scale)
Change in perceived stress from baseline | baseline, immediately post-intervention, 4 weeks post-intervention
  Change in Perceived stress scale from baseline
Change in migraine-related disability/impact from baseline | baseline, immediately post-intervention, 4 weeks post-intervention
  Change in migraine-related disability/impact from baseline(one month MIDAS and HIT-6)
Change in anxiety from baseline | baseline, immediately post-intervention, 4 weeks post-intervention
  Change in anxiety from baseline (state-trait anxiety measure)
Change in depression from baseline | baseline, immediately post-intervention, 4 weeks post-intervention
  Change in depression from baseline(PHQ-9)
Change in mindfulness from baseline | baseline, immediately post-intervention, 4 weeks post-intervention
  Change in mindfulness from baseline(Five facet mindfulness scale)
Qualitative interviews | immediately post-intervention
  Participants will be interviewed qualitatively
Change in migraine severity from baseline | baseline, immediately post-intervention, 4 weeks post-intervention
  Change in Migraine intensity (1-10) tracked via headache logs from baseline
Change in Migraine duration from baseline | baseline, immediately post-intervention, 4 weeks post-intervention
  Length of migraines (tracked via headache logs)
Change in quality of life from baseline | baseline, immediately post-intervention, 4 weeks post-intervention
  Change in Migraine specific quality of life from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca E Wells, MD, MPH, Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Wells RE, Burch R, Paulsen RH, Wayne PM, Houle TT, Loder E. Meditation for migraines: a pilot randomized controlled trial. Headache. 2014 Oct;54(9):1484-95. doi: 10.1111/head.12420. Epub 2014 Jul 18. PMID 25041058